CLINICAL TRIAL: NCT01154348
Title: A Phase 1b, Randomized, Placebo-Controlled Study to Assess the Safety and Pharmacokinetics of Double-Blind S-707106 Alone and in Combination With Open-Label Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Assess Safety and Pharmacokinetics of Double-Blind S-707106 Alone and in Combination With Open-Label Metformin in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1011N0913
Record Dates: First submitted 2010-06-25; First posted 2010-06-30 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — S-707106; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Washout period, S-707106 tablet (Experimental): 14-day washout of metformin, followed by S-707106 once daily for 14 days under fed conditions
  Interventions: Drug: S-707106
- Washout, placebo (Placebo Comparator): 14-day washout of metformin followed by placebo for S-707106 once daily for 14 days under fed conditions
  Interventions: Drug: Placebo
- Maintenance, S-707106 tablet plus metformin (Experimental): 14-day maintenance of metformin, followed by S-707106 once daily plus open-label metformin twice daily for 14 days under fed conditions
  Interventions: Drug: Metformin, S-707106 plus metformin
- Maintenance, placebo plus metformin (Placebo Comparator): 14-day maintenance of metformin, followed by placebo for S-707106 once daily plus open-label metformin twice daily for 14 days under fed conditions
  Interventions: Drug: Metformin, placebo plus metformin

INTERVENTIONS:
Drug: S-707106 — Tablet, taken once daily with morning meal
  Arms: Washout period, S-707106 tablet
Drug: Placebo — Placebo tablet, taken once daily with morning meal
  Arms: Washout, placebo
Drug: Metformin, S-707106 plus metformin — Metformin twice daily maintenance, S-707106 tablet taken once daily with morning meal with metformin dosed twice daily
  Arms: Maintenance, S-707106 tablet plus metformin
Drug: Metformin, placebo plus metformin — Metformin twice daily maintenance, placebo tablet taken once daily with morning meal with metformin twice daily
  Arms: Maintenance, placebo plus metformin

SUMMARY:
The purpose of this study is to determine the safety and pharmacokinetics of double-blind S-707106 alone and in combination with open-label metformin in patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
Safety will be evaluated by monitoring of treatment-emergent adverse events, clinical laboratory evaluations, vital signs, 12-lead electrocardiograms, 24-hour telemetry monitoring, and physical exams. Specific study withdrawal criteria during washout periods of metformin have been established for loss of glycemic control, i.e., glucose monitoring. Pharmacokinetic assessments of monotherapy cohort versus add-on therapy will be performed

ELIGIBILITY:
Inclusion Criteria:

* Body mass index range (25.0-38 kg/m2) with type 2 diabetes mellitus receiving stable dose of metformin BID for the previous 60 days for glucose control
* Patients sterile or agree to use approved method of contraception
* No clinically significant abnormal tests
* Hemoglobin A1c level ≤10.5%

Exclusion Criteria:

* History of clinical manifestations of significant metabolic, hepatic, renal, and hematological pulmonary, cardiovascular, gastrointestinal, urological, neurological, or psychiatric disorders other than type 2 diabetes mellitus
* Uncontrolled diabetes
* Exclusionary labs - fasting blood sugar, low hemoglobin, elevated liver function tests, positive result for human immunodeficiency virus, hepatitis B surface antigen, and anti-hepatitis C virus
* Low creatinine clearance
* History of myocardial infarction within past 90 days or other cardiovascular conditions
* Prior exposure to S-707106
* Treatment with investigational study drug within 30 days of study admission day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics of multiple-dose oral administration of S-707106 in fed state in patients with type 2 diabetes mellitus | Adverse events will be monitored from the time of informed consent through 28 days after the last dose of study treatment. Samples for S-707106 will be collected on Days 1, 7, 10, 12, 13, and 14
  Safety will be evaluated by monitoring of treatment-emergent adverse events, clinical laboratory evaluations, vital signs, 12-lead electrocardiograms, 24-hour telemetry monitoring and physical exams. Pharmacokinetic evaluation of monotherapy cohort versus add-on therapy will be done
Safety and pharmacokinetics of multiple-dose oral co-administration of S-707106 and metformin in fed state in patients with type 2 diabetes mellitus | Adverse events will be monitored from the time of informed consent through 28 days after the last dose of study treatment. Samples for S-707106 collected on Days 7, 10, 12, 13, and 14. Samples for metformin collected on Days -1, 7, 10, 12, 13, and 14
  Safety will be evaluated by monitoring of treatment-emergent adverse events, clinical laboratory evaluations, vital signs, 12-lead electrocardiograms, 24-hour telemetry monitoring and physical exams. Pharmacokinetic evalaution of monotherapy cohort versus add-on therapy will be done

SECONDARY OUTCOMES:
The effect of multiple doses of S-707106 on pharmacokinetics of metformin | On Day 14 and on day prior to initiation of dosing of S-707106
The effect of multiple doses of metformin on pharmacokinetics of S-707106 | On Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Dennis Ruff, MD, San Antonio, Texas, United States